CLINICAL TRIAL: NCT05915273
Title: Relapse and Failure Rates Between CAD/CAM and Conventional Fixed Retainers: A 2-year Follow-up of a Randomized Controlled Clinical Trial
Brief Title: Relapse and Failure Rates Between CAD/CAM and Conventional Fixed Retainers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32524
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAD/CAM group (Experimental)
  Interventions: Other: Computer Aided Design/ Computer Aided Manufacturing Retainers
- Lab group (Active Comparator)
  Interventions: Other: Lab-based Retainers
- Chairside group (Active Comparator)
  Interventions: Other: Chairside Retainers

INTERVENTIONS:
Other: Computer Aided Design/ Computer Aided Manufacturing Retainers — Custom-bent fixed retainer wires from an in-office CAD/CAM system with FixR software and the BenderI machine (YOAT Corporation, Lynwood, WA). Dentaflex wires- round, 0.5mm in diameter, three-stranded Stainless Steel (Dentaurum GmbH & Co., Ispringen, Germany)- were used for the CAD/CAM group
  Other Names: CAD/CAM
  Arms: CAD/CAM group
Other: Lab-based Retainers — The lab group used the same type of wire as the CAD/CAM group but was manually bent by a lab technician
  Arms: Lab group
Other: Chairside Retainers — The chairside group used three-stranded Stainless Steel, 0.974mm x 0.402 mm, flexible Ortho-FlexTech wires (Reliance, Itasca, IL)
  Arms: Chairside group

SUMMARY:
The aim of this study was to compare the differences in relapse and failure rates in patients treated with fixed retainers (FRs) using Computer-Aided Design/Computer-Aided Manufacturing technology, lab-based technique, and chairside method.

ELIGIBILITY:
Inclusion Criteria:

* completion of comprehensive orthodontic treatment
* class I molar and canine relationships
* indication for a fixed retainer on the mandibular anterior teeth.
* no extractions done as part of their treatment.
* Treatment with preadjusted edgewise appliance.

Exclusion Criteria:

* refusal to participate
* refusal to have fixed retainers
* poor oral hygiene
* non-compliance

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in intercanine width (ICW) | 2 years
  ICW was measured on the Meshlab software using the 3D ruler measurement tool. Pre-treatment, post-treatment, and post-retention measures were recorded and any change in the ICW was considered relapse.
Change in Little's Irregularity Index (LII) | 2 years
  ICW was measured on the Meshlab software using the 3D ruler measurement tool. Pre-treatment, post-treatment, and post-retention measures were recorded and any change in the LII was considered relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Giau Tran, Principal Investigator — Department of Orthodontics, Saint Louis University, Saint Louis, MO, USA.; Ryan Rucker, Principal Investigator — Department of Orthodontics, Saint Louis University, Saint Louis, MO, USA.; Patrick Foley, PhD, Study Chair — Department of Orthodontics, Saint Louis University, Saint Louis, MO, USA.; Brent Bankhead, Study Chair — Department of Orthodontics, Saint Louis University, Saint Louis, MO, USA.; Samar M Adel, PhD, Study Director — Alexandria University; Ki B Kim, Study Director — Department of Orthodontics, Saint Louis University, Saint Louis, MO, USA.
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Tran G, Rucker R, Foley P, Bankhead B, Adel SM, Kim KB. Relapse and failure rates between CAD/CAM and conventional fixed retainers: a 2-year follow-up of a randomized controlled clinical trial. Eur J Orthod. 2024 Jan 1;46(1):cjad079. doi: 10.1093/ejo/cjad079. PMID 38168815